CLINICAL TRIAL: NCT00041093
Title: A Phase II Evaluation Of Docetaxel (NSC #628503) In The Treatment Of Persistent Or Recurrent Squamous Cell Carcinoma Of The Cervix
Brief Title: Docetaxel in Treating Patients With Persistent or Recurrent Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0127S; NCI-2012-02476 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000069442; GOG-0127S (Other: Gynecologic Oncology Group); GOG-0127S (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Cervical Squamous Cell Carcinoma, Not Otherwise Specified; Recurrent Cervical Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Docetaxel

ARMS (1):
- Treatment (docetaxel) (Experimental): Patients receive docetaxel IV over 1 hour on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate

SUMMARY:
Phase II trial to study the effectiveness of docetaxel in treating patients who have persistent or recurrent cervical cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the antitumor activity of docetaxel in patients with persistent or recurrent squamous cell carcinoma of the cervix.

II. Determine the toxicity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive docetaxel IV over 1 hour on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed persistent or recurrent squamous cell carcinoma of the cervix
* Progressive disease
* At least 1 unidimensionally measurable target lesion

  * At least 20 mm by conventional techniques
  * At least 10 mm by spiral CT scan
  * Tumors within a previously irradiated field are not considered target lesions
* One prior systemic chemotherapeutic regimen for advanced, metastatic, or recurrent squamous cell carcinoma of the cervix required

  * Chemotherapy administered as a radiosensitizer in conjunction with primary radiotherapy is not considered a systemic chemotherapy regimen
* Ineligible for a higher priority GOG protocol (e.g., any active Phase III GOG protocol or GOG-0076)
* Performance status - GOG 0-2
* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* Creatinine no greater than 1.5 times ULN
* No congestive heart failure
* No unstable angina, myocardial infarction, or new cardiac arrhythmia within the past 6 months
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection requiring antibiotics
* No greater than grade 1 sensory and motor neuropathy
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* At least 3 weeks since prior biologic or immunologic therapy directed at malignant tumor
* One prior noncytotoxic regimen (e.g., monoclonal antibodies, cytokines, or small-molecule signal transduction inhibitors) for recurrent or persistent disease allowed
* Recovered from prior chemotherapy
* No prior docetaxel
* No more than 1 prior cytotoxic chemotherapy regimen
* At least one week since prior hormonal therapy directed at malignant tumor
* Concurrent hormone replacement therapy allowed
* Recovered from prior radiotherapy
* Recovered from recent prior surgery
* At least 3 weeks since any prior therapy directed at malignant tumor
* No prior anticancer therapy that would preclude study
* No concurrent amifostine or other protective agents

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2002-06; Primary Completion 2006-10-23 (Actual)

PRIMARY OUTCOMES:
Duration of progression-free interval | 5 years
Frequency and duration of objective response as assessed on radiologic scan | 5 years
Frequency and severity of observed adverse effects | 5 years
Survival time | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Agustin Garcia, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States